CLINICAL TRIAL: NCT02949817
Title: The Effect of Digital Rehabilitation System With Wearable Multi-IMU (Inertial Measurement Unit) Sensors on Upper Limb Functions in Children With Brain Injury: Single Blind Randomized Controlled Study
Brief Title: The Effect of Digital Rehabilitation System With Wearable Multi-IMU (Inertial Measurement Unit) Sensors on Upper Limb Functions in Children With Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-2015-0097
Record Dates: First submitted 2016-03-14; First posted 2016-10-31 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Cerebral Palsy; Children With Brain Injury
Keywords: upper limb function; multi-IMU (inertial measurement unit) sensors; Melbourne Assessment of Unilateral Upper Limb Function (MUUL-2)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMU sensor training group(intervention group) (Experimental): video-game based rehabilitation therapy system training group
  Interventions: Device: digital rehabilitation system with wearable multi-IMU(inertial measurement unit) sensors (Rapael kids)
- Conventional OT group (control group) (Active Comparator): conventional training group (control group)
  Interventions: Other: Conventional OT group

INTERVENTIONS:
Device: digital rehabilitation system with wearable multi-IMU(inertial measurement unit) sensors (Rapael kids) — 1.The Rapael kids, a video-game based rehabilitation therapy system using IMU sensors as a game interface, newly-developed in Korea will be used on upper limb function of children with pediatric brain injury patients. 20 of All 40 children will receive the conventional occupational therapy and additional video-game based rehabilitation therapy, 30 minutes daily 5 times per week, for 4 weeks.
  Arms: IMU sensor training group(intervention group)
Other: Conventional OT group — 2. Conventional OT group will recieve the conventional occupational therapy and one more conventional occupational therapy additionally. The additional occupational therapy training will be performed 30 minutes daily 5 times per week, for 4 weeks.
  Arms: Conventional OT group (control group)

SUMMARY:
This study was designed to establish the clinical evidence for effect of video-game based rehabilitation therapy system using IMU sensors as a game interface, newly-developed in Korea, on upper limb function of children with cerebral palsy. First, the investigators would compare the effect of video-game based rehabilitation therapy to conventional occupational therapy.

DETAILED DESCRIPTION:
* Purpose: to elucidate the effect of video-game based rehabilitation therapy system on upper limb function of children with cerebral palsy compared to conventional occupational therapy
* Subjects: total 30 children with cerebral palsy whose upper limb functions are impaired (all 30 children will receive the conventional occupational therapy, but 15 of these children will receive the additional video-game based rehabilitation therapy)
* Intervention: 4 weeks of therapy (6 days per week)
* Studies: functional MRI, computerized motion analysis, upper limb functional assessment (MUUL, ULPRS), ADL evaluation, cognitive evaluation
* Evaluation plan: 1) pre-intervention, 2) post-4 weeks of intervention, 3) 8 weeks after end of intervention

ELIGIBILITY:
Inclusion Criteria:

* MACS (Manual ability classification system) level I, II, III, IV
* Patients without cognitive impairment who are able to comply with protocol-required procedure
* male or female, 4 to 18 years

Exclusion Criteria:

* Patients with cognitive impairment who are unable to comply with protocol-required procedure
* Patients with significant visual impairment
* Patients with presence or history of musculoskeletal anomaly who are unable to apply device

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Total score of Melbourne Assessment of Unilateral Upper Limb Function | 8 weeks
  MUUL is the test of unilateral upper limb function is a validated and reliable tool for evaluating quality of upper limb movement in children with neurological conditions. It comprises 14 test items of reaching to, grasping, releasing and manipulating simple objects. Scoring is completed for the 30 item scores using a three, four or five point scale and the individually defined scoring criteria. The test will be done by occupational therapist. The total score of MUUL will be used for analysis.

SECONDARY OUTCOMES:
Total score of upper limb physician's rating scale (ULPRS) | 8 week
  ULPRS assess changes in the movement pattern, focusing on all 3 levels of the arm (palm, forearm, and elbow) to determine whether there is an isolated functional impairment, such as thumb in palm, restricted forearm supination, or a total flexion pattern with thumb in palm, wrist in flexion, forearm supinated, and elbow flexed. The score sheet includes 9 items, and 3-, 4-, and 5-point scales are used to score each component of movement tested. The total score of ULPRS will be used for analysis.
Scaled scores of Pediatric Evaluation of Disability Inventory (PEDI-selfcare) | 8 week
  PEDI is a descriptive measure of a child's current functional performance. It measures both capability and performance of functional activities in three content domains: Self-care, Mobility, Social function. PEDI-selfcare section will be administered by occupational therapist. The Scaled scores of PEDI-selfcare will be used for analysis.
Kinematic data of computerized 3D motion analysis | 8 week
  3D motion analysis will be performed using a computerized motion analysis system (VICON MX-T10 System with 6 infrared cameras, Oxford Metrics Inc., Oxford, UK) to measure the kinematic data (angle of each joint) during the task of drinking from a cup. Kinematic data of forearm pronation or supination, wrist flexion or extension, ulnar deviation or radial deviation will be used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No